CLINICAL TRIAL: NCT05093946
Title: Psychometric Measurement Properties of the German Version of the Michigan Hand Questionnaire in Patients After Flexor Tendon Repair
Brief Title: Psychometric Measurement Properties of the Michigan Hand Questionnaire in Patients After Flexor Tendon Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00929a
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Flexor Tendon Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate the psychometric properties of the German Version of the Michigan Hand Questionnaire in patients with flexor tendon injuries, including reliability, validity and interpretability.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* ≥ 18 years old
* Understanding of the German language (written and oral)
* Single and multiple finger injuries
* Primary flexor tendon injuries in Zone I-V for the fingers and/ or thumb
* Treated by the hand surgery department at the Inselspital Bern
* Treated with at least a 4-strand core suture

Exclusion Criteria:

* < 18 years old
* Inability to follow the procedures of the study, e.g. due to language problems, diagnosed psychological disorders or dementia of the patients
* Replantation of the injured finger
* Fracture of the injured finger
* Primary tendon reconstructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with flexor tendon injuries in Zone I-V for in the fingers and/or thumb.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Michigan Hand Questionnaire (MHQ) | 6, 13, 13 1/2 and 26 weeks after tendon repair
  The MHQ is a hand specific questionnaire used to measure the ability in daily function. The total score ranges from 0 to 100, with higher scores indicating better performance.

SECONDARY OUTCOMES:
Disabilities of Shoulder, Arm and Hand Questionnaire | 6, 13 and 26 weeks after tendon repair]
  The DASH questionnaire is a region-specific outcome instrument. The patient will rate 30-items about disability or symptoms by rating the degree of difficulty in doing various activities. The scores of all items are used to calculate a score ranging from 0 (no disability) to 100 (most severe disability). The DASH is a region-specific outcome instrument. The patient will rate 30-items about disability or symptoms by rating the degree of difficulty in doing various activities. The scores of all items are used to calculate a score ranging from 0 (no disability) to 100 (most severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Tobler, Dr. phil., Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No